CLINICAL TRIAL: NCT05297344
Title: Clinical Study of the Direct Pulp Capping in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, JINjin Yu, Attending Physicians, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHZhejiangU-2022（22）
Record Dates: First submitted 2022-03-14; First posted 2022-03-28 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Direct Pulp Capping; Pulpotomy; Primary Teeth
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct pulp capping (Experimental): If a pulp exposure occurred, direct pulp capping will be performed according to the parents' wishes
  Interventions: Procedure: direct pulp capping
- pulpotomy (Active Comparator): If a pulp exposure occurred, pulpotomy will be performed according to the parents' wishes
  Interventions: Procedure: pulpotomy

INTERVENTIONS:
Procedure: direct pulp capping — direct pulp capping
  Arms: direct pulp capping
Procedure: pulpotomy — pulpotomy
  Arms: pulpotomy

SUMMARY:
Research content: select the patients with accidental pulp exposure or decayed pulp exposure in the pediatric dentistry department of The Affiliated Stomatology Hospital of Zhejiang University School of Medicine from February 2022 to October 2022.

1. Strictly implement the case selection criteria to reduce the deviation. 2. Conduct uniform training and assessment for doctors. 3. Record in detail: the age, gender, tooth position, cavity type, x-Ray examination, size and reason of pulp exposure, time of hemostasis, filling material, signs and symptoms of initial consultation and follow-up, etc. 4. Analyze the clinical data to study the success rate of direct pulp capping of primary teeth; analyze the influence of various factors to study how to improve the success rate of direct pulp capping of primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* No irreversible signs or symptoms of pulpitis in the affected tooth.
* Mechanical pulp exposure caused by cavity preparation or trauma, or pulp exposure after decayed tissue removal, with healthy dentin around the pulp exposure.
* The size of the exposed pulp<1 mm.
* The morphology of pulp tissue at the pulp exposure is normal, and the bleeding should be able to be controlled within 5 minutes.
* X-ray showed that there was no abnormal resorption or fracture of the root and no lesions around the root.

Exclusion Criteria:

* The child is unable to cooperate with the treatment.
* Pulp exposure > 1 mm.
* Irreversible signs or symptoms of pulpitis in the affected tooth.
* Abnormal morphology of the pulp tissue at the pulp exposure, much bleeding and inability to stop bleeding.
* X-ray shows: abnormal resorption or fracture of the tooth root and lesions around the root.
* The parents or the child refused to participate in the experiment.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Success rate of the direct pulp capping | 12 months
  The success rate of the direct pulp capping of primary teeth

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Stomatology, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No